CLINICAL TRIAL: NCT06783959
Title: Deconstructing Fast-Food Consumption Among Female University Students
Brief Title: Deconstructing Fast-Food Consumption Among Female University Students University Women
Acronym: Fast Food
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Fast Food University Women
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Identities; Fast Food Consumption; University Female Student

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant Selection: female students aged 18-24 from Mansoura University, with a focus on students from two practical faculties (Faculty of Science and Faculty of Agriculture) and two theoretical faculties (Faculty of Education and Faculty of Arts).

SUMMARY:
This study aims to explore the relationship between fast food consumption and identity formation among adolescent female university students, examining how their dietary choices reflect and shape their self-perceptions.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between fast food consumption and identity formation among adolescent female university students, with a specific focus on how their dietary choices reflect and shape their self-perceptions. Key research questions include understanding the factors that drive fast food consumption, exploring how these choices influence self-identity, and examining the role of social and cultural dynamics in shaping dietary behavior. The study also seeks to highlight the role of nurses in communicating nutritional knowledge and supporting adolescents in developing healthier eating habits. By examining the psychosocial drivers behind fast food consumption, this research aims to inform public health initiatives and health education strategies that are attuned to the needs and identities of university students.

The findings from this study are expected to contribute valuable insights into the relationship between food choices and identity among adolescent women, providing a foundation for health interventions that consider both the social and personal aspects of dietary behavior. Understanding that food choices are intertwined with self-concept, social belonging, and cultural trends can help public health professionals and nurses develop targeted strategies that resonate with the lived experiences of young women. By addressing these factors, universities can implement health policies and education programs that not only encourage healthier dietary habits but also respect and support the identity development of adolescent female students. Ultimately, this research underscores the importance of a holistic approach to health education, where nurses and other healthcare professionals play a proactive role in guiding adolescents toward healthier lifestyle choices in a way that is meaningful, sustainable, and aligned with their values.

ELIGIBILITY:
Inclusion Criteria:

1. Female students.
2. Aged between 18 and 24 years,
3. Currently enrolled as a student at Mansoura University
4. Students from all grades (1 to 5) within the selected faculties.
5. accept to provide written informed consent to participate in the study

Exclusion Criteria:

1. Male students.
2. outside the age range of 18 to 24 years.
3. medical conditions that significantly affect dietary choices or
4. eating behaviors disorder
5. eating disorders,
6. metabolic disorders
7. specific dietary regimens prescribed by healthcare professionals.
8. previously participated in this study or similar research

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be conducted at Mansoura University in Egypt, targeting four faculties: two practical faculties (Faculty of Science and Faculty of Agriculture) and two theoretical faculties (Faculty of Education and Faculty of Arts). This selection allows for diverse perspectives, with students pursuing both scientific and theoretical fields, which may influence their attitudes toward dietary choices and identity. The study will include adolescent female students from grades 1 to 5 across the selected faculties, ensuring a representative sample of different ages and stages of academic progression.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Knowledge of fast food consumption: | 3 months
  included 14 items to measure students' knowledge about fast food, side effects, and proper and healthy nutrition
  Scoring system:
  The score of each item varied from 0 to 2. The minimum and maximum score for the knowledge subscale was 0 and 28, respectively
Attitude towards fast food consumption | 3 months
  The scores will be graded based on five-point the Likert scale (from strongly agree to strongly disagree) or (from very important to not at all important), and the score of each item varied from 1 to 5. The minimum and maximum score for the attitude subscale was 14 and 350, respectively.
Perceived Behavioral Control | 3 month
  was measured by 18 indirect items (9 items of control beliefs, 9 items of perceive power) Scoring system The tool will be scored based on five-point the Likert scale (from strongly agree to strongly disagree) or (from extremely difficult to extremely easy), and the score of each item varied from 1 to 5.
Subjective norms | 3 month
  measured by 10 indirect items (5 items of normative beliefs, 5 items of motivation to comply) Scoring system The too; was be scored based on five-point the Likert scale (from strongly agree to strongly disagree) or (from very important to not at all important), and the score of each item varied from 1 to 5. The minimum and maximum score for the subjective norm subscale was 5 and 125, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr/ Basma Wageah Mohamed Mohamed Elrefay, Al Mansurah, Dakahlia Governorate, Egypt